CLINICAL TRIAL: NCT06540664
Title: Evaluating Efficacy and Safety of Auricular Acupuncture in Treating Insomnia Post-stroke: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Auricular Acupuncture in Treating Insomnia Post-stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, NGUYEN THI THUY AN, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1100/HDDD-DHYD
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Insomnia, Secondary; Post-stroke Depression
Keywords: insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular Acupuncture (Experimental): Participants received Auricular Acupuncture every 5 days for 2 weeks combined with sleep hygiene, then stopped acupuncture and monitored for effectiveness after 4 weeks.
  Interventions: Other: Auricular Acupuncture needles
- Sham Auricular Acupuncture (Sham Comparator): Participants received sham Auricular Acupuncture every 5 days for 2 weeks combined with sleep hygiene, then stopped acupuncture and monitored for effectiveness after 4 weeks.
  Interventions: Other: Sham Auricular Acupuncture needles

INTERVENTIONS:
Other: Auricular Acupuncture needles — Auricular Acupuncture needles 5 days in 2 weeks
  Arms: Auricular Acupuncture
Other: Sham Auricular Acupuncture needles — Sham Auricular Acupuncture needles 5 days in 2 weeks
  Arms: Sham Auricular Acupuncture

SUMMARY:
The goal of this clinical trial is to learn if Auricular acupuncture works to treat Insomnia Post-stroke patients. It will also learn about the safety of Auricular. The main questions it aims to answer are:

* Does Auricular acupuncture reduce the time it took participants to fall asleep?
* Dose Auricular acupuncture increase the number of hours participants slept?
* Dose Auricular acupuncture improve sleep quality as measured by The Pittsburgh Sleep Quality Index (PSQI)?
* What medical problems do participants have when taking Auricular acupuncture? Researchers will compare Auricular acupuncture to a sham Auricular acupuncture (a look-alike acupuncture needles that contains no needles) to see if Auricular acupuncture works to treat insomnia post-stroke.

Participants will:

* Take Auricular acupuncture or sham Auricular acupuncture every 5 days for 4 weeks.
* Checkups and evaluate sleep onset time, sleep hours, and sleep quality every 5 days for 4 weeks.
* Keep a diary sleep of their symptoms and the number of times they use sleeping pills.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, with a post-stroke period of 03 months or more, based on discharge papers or medical records.
* Patients who meet the diagnostic criteria for insomnia according to the DSM-V of the American Psychiatric Association for at least 3 months.

Exclusion Criteria:

* Patients with insomnia before the stroke.
* Patients diagnosed with other sleep disorders such as sleep apnea syndrome, narcolepsy.
* Patients diagnosed with neurological diseases or psychiatric disorders such as: Anxiety disorders, autism spectrum disorders, depression, obsessive-compulsive disorder, behavioral disorders affecting sleep before the stroke.
* Patients are using antidepressants, psychiatric drugs.
* Patients participating in other clinical trials with behavioral, psychological or complementary medical interventions during the study period.
* Patients not cooperating during data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change sleep quality as measured by The Pittsburgh Sleep Quality Index (PSQI) | Baseline and Week 4
  The Pittsburgh Sleep Quality Index (PSQI) is a validated, self-reported instrument assessing sleep quality over 1 month. Possible scores range from 0 to 21. PSQI < 5 (good sleep quality), PSQI >5 (poor sleep quality)

SECONDARY OUTCOMES:
Change number of hours slept as measured by The Pittsburgh Sleep Quality Index (PSQI) | Baseline and Week 4
  The Pittsburgh Sleep Quality Index (PSQI) is a validated, self-reported instrument assessing sleep quality over 1 month. The score of hours slept range 0 (hours of sleep > 7 hours) to 3 (Hours of sleep < 4 hours)
Change the time it took participants to fall asleep as measured by The Pittsburgh Sleep Quality Index (PSQI) | Baseline and Week 4
  The Pittsburgh Sleep Quality Index (PSQI) is a validated, self-reported instrument assessing sleep quality over 1 month. The score of time it took participants to fall asleep range 0 (<15 minutes) to 3 ( >60 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- HoChiMinh University of Medicine and Phamacy, Ho Chi Minh City, Vietnam